CLINICAL TRIAL: NCT02098408
Title: A Randomised Clinical Trial Examining Cognitive Remediation Plus Standard Treatment Versus Standard Treatment in Participants at Ultra-High Risk of Psychosis. - Effect on Cognitive Functioning, Functional Outcome and Symptomatology.
Brief Title: Effects of Neurocognitive and Social Cognitive Remediation in Patients at Ultra-High Risk of Psychosis
Acronym: FOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Center for Clinical Intervention and Neuropsychiatric Schizophrenia Research, CINS (Unknown); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-6-2013-015
Record Dates: First submitted 2014-03-18; First posted 2014-03-28 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-03

CONDITIONS: Patients at Ultra-high Risk of Psychosis
Keywords: Ultra-high risk psychosis; Schizophrenia prodrome; Cognitive remediation
MeSH Terms: interventions — Cognitive Remediation; Serum Bactericidal Test

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment + cognitive remediation (Experimental): The cognitive remediation therapy targets neurocognition as well as social cognition.
  Interventions: Behavioral: Cognitive remediation; Behavioral: Standard treatment
- Standard treatment (Active Comparator): Patients allocated to the control condition are free to choose whatever standard treatment they are offered by the clinicians managing their treatment. Usually standard treatment consists of regular contact to health professionals in the in- and outpatient facilities in Copenhagen, Denmark, and encompass different kinds of supportive counselling
  Interventions: Behavioral: Standard treatment

INTERVENTIONS:
Behavioral: Cognitive remediation — Neurocognition will be trained using the NEAR model (Medalia et al. 2003), whereas the training of social cognitive skills will be by use of the SCIT manual (Social Cognition and Interaction Training) developed by Roberts et al. 2014.
  The intervention consists of 24 group sessions taking place once a week (two hours) and additional neurocognitive training at home. Furthermore, there will be a total of 12 individual sessions aiming at bridging the cognitive training to the everyday functioning of the patients.
  Other Names: Neuropsychological & Educational Approach to Remediation (NEAR) using software from Scientific Brain Training Pro (SBT) and Posit Science.; Social Cognition and Interaction Training (SCIT)
  Arms: Standard treatment + cognitive remediation
Behavioral: Standard treatment — Patients allocated to the control condition are free to choose whatever standard treatment they are offered by the clinicians managing their treatment. Usually standard treatment consists of regular contact to health professionals in the in- and outpatient facilities in Copenhagen, Denmark, and encompass different kinds of supportive counselling.

SUMMARY:
Cognitive deficits are known to be a core feature of schizophrenia and seem to become manifest in the prodromal or Ultra-High Risk (UHR) state of psychosis. The cognitive deficits are known to pose a critical barrier to functional recovery. Hence it is of vital importance to find intervention strategies that can alleviate these cognitive deficits and consequently improve daily functioning, and quality of life, as well as the prognosis for UHR-patients. The investigators will examine whether:

* Cognitive remediation therapy will be superior to standard treatment in improving cognitive functioning in UHR- patients (null hypothesis: No difference between the two groups).
* Cognitive remediation therapy will be superior to standard treatment in improving psychosocial functioning and clinical symptoms in UHR-patients (null hypothesis: No difference between the two groups).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 yrs.
* Fulfill criteria for being at Ultra-High Risk of psychosis (defined by one or more of the following):

  * Vulnerability (Trait and State Risk Factor) Group: Individuals with a combination of a trait risk factor (schizotypal personality disorder or a family history of psychotic disorder in a first degree relative) and a significant deterioration in functioning, or sustained low functioning during the past year.
  * Attenuated Psychotic Symptoms (APS) Group: Individuals with sub-threshold (intensity or frequency) positive psychotic symptoms. The symptoms must have been present during the past year.
  * Brief Limited Intermittent Psychotic Symptoms Group (BLIPS): Individuals with a recent history of frank psychotic symptoms that resolved spontaneously (without antipsychotic medication) within one week. The symptoms must have been present during the past year.
* Provided informed consent.

Exclusion Criteria:

* Past history of a treated or untreated psychotic episode of one week's duration or longer
* Psychiatric symptoms that are explained by a physical illness with psychotropic effect or acute intoxication (e.g., cannabis use).
* Diagnosis of a serious developmental disorder, e.g,. Asperger's syndrome
* Currently receiving treatment with metylphenidate.
* Rejects providing informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Brief Assessment of Cognition in Schizophrenia (BACS) | 6 and 12 months
  BACS will be used to assess changes in cognition at the cessation of treatment at (6 months) and 12 months post baseline.

SECONDARY OUTCOMES:
Personal and Social Performance Scale (PSP) | 6 and 12 months
Brief Psychiatric Rating Scale Expanded Version (BPRS-E) | 6 and 12 months
Scale for the Assessment of Negative Symptoms (SANS) | 6 and 12 months
The Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 and 12 months

OTHER OUTCOMES:
Schizophrenia Prediction/Proneness Instrument - Adult Version (SPI-A) | 6 and 12 months
Behaviour Rating Inventory of Executive Function -Adult Version (BRIEF-A) | 6 and 12 months
Global Functioning: Social and Role Scales | 6 and 12 months
Quality Of Life Scale (QOLS). | 6 and 12 months
Comprehensive Assessment of At-Risk Mental States (CAARMS) | 6 and 12 months
The Awareness of Social Inference Test (TASIT) | 6 and 12 months
Emotion Recognition Task (ERT) | 6 and 12 months
  Emotion Recognition Task from CANTAB
Social Responsiveness Scale (SRS) | 6 and 12 months
Social Cognition Screening Questionnaire (SCSQ) | 6 and 12 months
Adverse events | 6 and 12 months
  Number of participants with adverse events
The High-Risk Social Challenge (HiSoC) Task | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, Professor, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital; Louise B Glenthøj, MsC, Study Director — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Kristensen TD, Ebdrup BH, Hjorthoj C, Mandl RCW, Raghava JM, Jepsen JRM, Fagerlund B, Glenthoj LB, Wenneberg C, Krakauer K, Pantelis C, Glenthoj BY, Nordentoft M. No Effects of Cognitive Remediation on Cerebral White Matter in Individuals at Ultra-High Risk for Psychosis-A Randomized Clinical Trial. Front Psychiatry. 2020 Aug 28;11:873. doi: 10.3389/fpsyt.2020.00873. eCollection 2020. PMID 33005161
- [Derived] Glenthoj LB, Mariegaard LS, Fagerlund B, Jepsen JRM, Kristensen TD, Wenneberg C, Krakauer K, Medalia A, Roberts DL, Hjorthoj C, Nordentoft M. Cognitive remediation plus standard treatment versus standard treatment alone for individuals at ultra-high risk of developing psychosis: Results of the FOCUS randomised clinical trial. Schizophr Res. 2020 Oct;224:151-158. doi: 10.1016/j.schres.2020.08.016. Epub 2020 Aug 29. PMID 32873460
- [Derived] Wenneberg C, Nordentoft M, Rostrup E, Glenthoj LB, Bojesen KB, Fagerlund B, Hjorthoj C, Krakauer K, Kristensen TD, Schwartz C, Edden RAE, Broberg BV, Glenthoj BY. Cerebral Glutamate and Gamma-Aminobutyric Acid Levels in Individuals at Ultra-high Risk for Psychosis and the Association With Clinical Symptoms and Cognition. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Jun;5(6):569-579. doi: 10.1016/j.bpsc.2019.12.005. Epub 2019 Dec 19. PMID 32008981
- [Derived] Glenthoj LB, Fagerlund B, Randers L, Hjorthoj CR, Wenneberg C, Krakauer K, Vosgerau A, Gluud C, Medalia A, Roberts DL, Nordentoft M. The FOCUS trial: cognitive remediation plus standard treatment versus standard treatment for patients at ultra-high risk for psychosis: study protocol for a randomised controlled trial. Trials. 2015 Jan 27;16:25. doi: 10.1186/s13063-014-0542-8. PMID 25623736